CLINICAL TRIAL: NCT03885206
Title: Effectiveness and Clinical Outcomes of Municipal Acute Wards Versus a General Hospital: a Multicenter, Randomized Controlled Trial
Brief Title: Effectiveness and Clinical Outcomes of Municipal Acute Wards Versus a General Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: Extrastiftelsen, Akersgatab28, No-0158Oslo, Norway (Other Government); The National Association for Heart and Lung Disease, Jessheim, Norway (Other); University of Oslo (Other); University Hospital, Akershus (Other); Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Ann-Chatrin Leonardsen, Associate Professor, Ostfold University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS2522-40480
Record Dates: First submitted 2018-12-05; First posted 2019-03-21 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Patient Experience; Medical Emergencies; Mortality; Morbidity; Co-morbidity; Quality of Life

STUDY DESIGN:
Intervention Model Description: The referring physician in a casualty in the casualty will judge the patients´ eligibility for inclusion, Study nurses in the casualty will invite participants, and receive patients´ written informed consent to participate, and then randomize the patients to either the MAW or the hospital, using a simple randomization procedure with numbered sheets in sealed, opaque envelopes. The patients will then be transported to the MAW or hospital according to the random allocation procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital (Experimental): Level of healthcare service: Patients who can be admitted to a municipal acute ward (MAW) will be admitted to the hospital instead, so that the intervention is that patients are admitted to a higher level facility than needed. Recieve medical treatment as usual.
  Interventions: Other: Level of healthcare services
- Municipal acute ward (No Intervention): Patients admitted to decentralized, municipal acute care wards after being assessed by a referring physician.

INTERVENTIONS:
Other: Level of healthcare services — Patiens judged to be eligible for admittance to a municipal acute care wrad will be admitted to hospital as an intervnetion, to be able to compare same patient groups.
  Arms: Hospital

SUMMARY:
Demographic changes in the industrialized world are expected to prompt a need for better organized and more efficient health care services. In order to curb costs, health care providers in many countries are searching for viable alternatives to hospitalizations. Norwegian white papers and reform documents presume that the municipalities will play a central role in meeting the growth in demand for health services. Central public policy documents and national research strategies highlight that we need pathways characterized by good quality and safe care, and which are responsive to needs, based on user involvement, continuity of care and successful collaboration within and between service levels. The 2012 Coordination Reform placed new responsibilities on municipalities in the delivery of primary health care services and on hospitals as deliverers of specialist services, as well as on the integration and collaboration between the two organizational levels. This reform mandates that all 428 Norwegian municipalities are obliged to establish or co-operate on establishing Municipal Acute Wards (MAW) (In Norwegian: Kommunale akutte døgnplasser), so as to alleviate pressure on hospitals. However, the research basis for these units is relatively weak. Hence, there is little information on the outcomes regarding the quality, cost-effectiveness, patient-reported as well as personnel-reported outcomes of this new level of care.

This study aims at assessing the outcome of admissions to MAWs compared to a general hospital for patients in need of acute care, that can be treated at a lower and decentralized level of health care, with potentially less resources than traditional hospitalizations. The study will use a Randomized Controlled Trial (RCT) design. It builds on previous research and systematic reviews, and aims to assess several outcomes, patient experiences (NORPEQ), health-related quality of life, short-term mortality and morbidity, and draws on linkages to national registers. The primary hypothesis is that there is no difference in patient experiences between admissions to a MAW versus a hospital. The secondary hypothesis was that there is no difference in outcomes such as readmission, length of stay, self-assessed health-related quality of life (HRQoL) measured by the EuroQol 5 items 5 level (EQ-5D-5L) index, and health status measured by the RAND-12, between patients admitted to a MAW versus a hospital

DETAILED DESCRIPTION:
No other randomized, controlled studies have been conducted to compare healthcare services as offered in MAWs to those offered in hospital. The study will use an RCT design, which is a strong study design. The study includes measures of patient experiences and HRQoL. The project is interdisciplinary and cross-sectoral, and it represents research in, about and with support from the municipalities, which is a prioritized area of research, together with health services research, for the owners of the Østfold Hospital Trust, Helse Sør-Øst (HSØ). The project incorporates users in the planning of the project, which may contribute better acceptance of and a successful completion of the project. This proposal addresses key aspects of the CR and other national strategic documents. The CR has mandated the establishment of MAWs all over Norway as of 2016, without any strong scientific documentation of cost-effectiveness. The study builds on data from previous research, stating that there is a need for more solid documentation about new levels of acute hospital care. The proposed study will assess several aspects of quality of care and will contribute useful information for evaluation and future planning of MAWs, as an alternative to hospitalization. Therefore the researchers think this project is timely. The MAWs in Østfold County are small to medium-sized and are expected to be representative for the majority of MAWs in Norway, and therefore of broad national interest. These outputs will be important for authorities, politicians, healthcare leaders, and professionals as well as researchers involved in developing, implementing and refining decentralized acute health care services as an alternative to hospitalization- to the best of the patients. Moreover, the project outputs will be of international interest, in particular in countries with national health insurance with broad coverage, as in the Nordic countries, the UK, Canada and Australia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to provide written, informed consent
* Eligible for admission at a MAW according to established admission criteria
* Assessed and referred by a GP, by a physician at the local Casualty (Legevaktslege), or a physician in a nursing home on the same day

Exclusion Criteria:

* Psychiatric or cognitive impairment
* No Norwegian national identification number
* Acute disability in elderly, requiring extensive diagnostic procedures
* Patients admitted to the MAW via the diagnostic loop*
* Previous admission to a MAW during the project period (to prevent patients being included more than once in the project)
* Insufficient Norwegian language skills to respond to the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sütterlin, Professor, Study Chair — Ostfold University College
Locations (1):
- Ostfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hospital | Municipal Acute Ward
Started | 49 | 115
Completed | 26 | 70
Not Completed | 23 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hospital | Municipal Acute Ward | Total
Number analyzed (Participants) | 49 | 115 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (19.9) | 70.7 (20.6) | 69.6 (20.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 77 | 106
  Male | 20 | 38 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
EQ-5D index [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D-3L is a generic measure of health status that provides a simple descriptive profile and a single index value. An EQ-5D summary index is derived by applying a formula that essentially attaches values to each of the levels in each dimension. The EQ-5D index utility score ranges from 0 to 1, where 0 indicates a worse health scenario and 1 indicates the best health scenario. The EQ VAS ranges from 0 to 100, where 0 represents the worst possible self-assessed health-related quality of life and 100 the best possible.
  units on a scale | 0.3 (0.4) | 0.3 (0.4) | 0.3 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Patient Experiences, NORPEQ
Description: Norwegian Patient Experience Questionnaire. Six of the eight NORPEQ items sum to produce an overall scale from 0 to 100, where 100 is the best possible experience of care. If respondents had missing values on more than half of the items, mean scores will be imputed.
Time Frame: 2-4 weeks after discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hospital | Municipal Acute Ward
Number analyzed (Participants) | 49 | 115
units on a scale | 78.7 (15.5) | 80.9 (9.8)

2. Secondary Outcome: 30-day Mortality
Description: Number of deaths within 30 days after discharge, all causes
Time Frame: 30 days
Reporting Status: Not Posted

3. Secondary Outcome: 30-day Re-admission
Description: Number of re-admissions to hospital or MAW within 30 days after discharge, all causes
Time Frame: 30 days
Reporting Status: Not Posted

4. Secondary Outcome: Length of Stay
Description: Number of days patients are admitted to either hospital or MAW
Time Frame: 8 days
Reporting Status: Not Posted

5. Secondary Outcome: Number of Inpatients Stays
Description: Number of inpatient stays in a healthcare institution
Time Frame: 3 months
Reporting Status: Not Posted

6. Secondary Outcome: Transfer of Patients Between MAW and Hospital
Description: Number of patients transferred from MAW to hospital
Time Frame: 1,5 year
Reporting Status: Not Posted

7. Secondary Outcome: Patient Experiences
Description: As measured by the NORPEQ questionnaire. The questionnaire consist of eight items. The overall scale goes from 0 to 100, where 100 is the best possible experience of care.
  The
Time Frame: 4 weeks after discharge
Reporting Status: Not Posted

8. Secondary Outcome: Health Status as Assessed With the RAND-12 Instrument
Description: The RAND-12 health status inventory (aka SF-12) is a commonly used health status instrument, which was developed as part of the Medical outcomes study in the 1980s. It uses 12 items from the SF-36 and can be aggregated to a physical health component score and an mental health component score.
Time Frame: 4 weeks after discharge
Reporting Status: Not Posted

9. Secondary Outcome: Eq5D5L
Description: Health related quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement
Time Frame: 1,5 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Hospital | Municipal Acute Ward
All-Cause Mortality (participants affected / at risk) | 5/49 | 4/115
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/115
Other Adverse Events (participants affected / at risk) | 0/49 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03885206/Prot_SAP_000.pdf